CLINICAL TRIAL: NCT00724542
Title: Evaluation of Lifestyle and Therapeutic Intervention on Impaired Glucose Tolerance(IGT) in Patients With Coronary Heart Disease.
Brief Title: Evaluation of Intervention on Impaired Glucose Tolerance(IGT) in Patients With Coronary Heart Disease.
Acronym: EIIGETPCHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Collaborators: Takeda (Industry)
Responsible Party: Yong Huo, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2006BAI01A02-11
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Heart Disease; Impaired Glucose Tolerance
MeSH Terms: conditions — Coronary Disease; Glucose Intolerance | interventions — voglibose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Placebo with lifestyle intervention
- Drug (Experimental): Voglibose tablets with lifestyle intervention
  Interventions: Drug: Voglibose tablets

INTERVENTIONS:
Drug: Voglibose tablets — 0.2mg Tid
  Arms: Drug

SUMMARY:
The purpose of this study is to determine whether therapeutic intervention on impaired glucose tolerance in patients with coronary heart disease can decrease the incidence of new onset DM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary heart disease
* Impaired Glucose Tolerance

Exclusion Criteria:

* Age < 40yr or > 75yr
* Diabetes Mellitus
* Scr > 2.0 mg/dL（176 μmol/L）
* ALT or AST > 2.5 ULN
* Hb < 90g/L
* Heart Failure
* Infection
* Undergo other interventional clinical trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
TypeⅡDiabetes Mellitus | 2 years

SECONDARY OUTCOMES:
Occurrence of Cardiovascular Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wenhui Ding, Professor, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China